CLINICAL TRIAL: NCT06256003
Title: A Randomized, Controlled, Parallel-Group, Intervention Study to Assess At-Home, Digital Therapy for Treating Adult Participants Ages 18-50 Years Old With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Assessing Mobile Apps for Adult ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Think Now Incorporated (Industry)
Collaborators: University of California, Los Angeles (Other); University of California, Berkeley (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAC-II
Record Dates: First submitted 2024-02-04; First posted 2024-02-13 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UC-A (Active Comparator): UC-0A is a digital mobile app intervention that uses cognitive control skills for task performance. The intervention is used once a day, 5 days a week, for 7 weeks.
  Interventions: Device: UC-A
- UC-N (Active Comparator): UC-0N is a digital mobile app intervention that uses cog control skills for problem solving. The intervention is used once a day, 5 days a week, for 7 weeks.
  Interventions: Device: UC-N

INTERVENTIONS:
Device: UC-A — Mobile app digital therapy
  Arms: UC-A
Device: UC-N — Mobile app digital therapy
  Arms: UC-N

SUMMARY:
The purpose of this clinical trial is to evaluate the effects of mobile app digital therapies on cognitive function and symptoms in adults diagnosed with ADHD.

DETAILED DESCRIPTION:
The study is a randomized, parallel group, controlled trial of two mobile app digital therapies. The study will consist of initial screening tests and diagnostics to determine eligibility, followed by outcome measure testing and treatment. On Day 0, the Baseline visit will occur wherein the pre-treatment (baseline) assessments will be conducted on-site. The Treatment period (Day 1 to Day 49) will involve using the digital therapy at home. Midpoint (Day 25) assessments will be conducted on-site to assess key outcomes. Final Post-Treatment (Day 50) assessments will be conducted on-site to assess key outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The participant is aged 18-50 years at time of consent
* Fluent in English.
* Available for 2 contiguous months to participate in study, including 3 in-person visits to the university.
* Able to sit in a regular chair for 30 minutes in a small room for testing.
* Able to use a keyboard with both hands.
* Normal or corrected to normal vision and hearing.
* Have a smart Phone.
* Estimated Intelligence Quotient (IQ) > 80 as assessed by the Wechsler Abbreviated Scale Intelligence (WASI-II) Matrix Reasoning and Vocabulary subtests.
* Meet established Diagnostic and Statistical Manual of Mental Health-Fifth Edition (DSM-5-TR) presentation for ADHD predominantly inattentive or combined subtype with clinically significant levels of impairment, diagnosed by semi-structured clinical interview and the Adult ADHD Clinical Diagnostic Scale (ACDS).

Exclusion Criteria:

* History of diagnosis of childhood neurodevelopmental disorder including autism spectrum disorder and dyslexia, other than ADHD or those specifically allowed in the Allowed Disorders section.
* Lifetime history of DSM5 bipolar disorder, psychotic disorder, panic disorder, agoraphobia, obsessive compulsive disorder as assessed with the MINI International Neuropsychiatric Interview (MINI).
* Current DSM5 diagnosis of posttraumatic stress disorder, or Major Depressive Disorder or Major Depressive Episode via self-report or as assessed with the MINI.
* Current Persistent Depressive Disorder (Dysthymia) or Anxiety Disorder if not on allowed medication that has been at a stable dose for at least 8 weeks (if on allowed medication with stable dose for 8 weeks, then allow).
* Substance or Alcohol Use Disorder rated as moderate or severe, with symptoms ≥ 4, as assessed by the MINI, or self-report of a Substance/Alcohol Use Disorder (allow endorsement of substance or alcohol use that does not meet moderate-severe use disorder criterion, if clean at visit).
* History of severe sleep disorder, narcolepsy, epilepsy/seizure disorder, brain tumor, stroke, TBI, severe concussion resulting in loss of consciousness and hospitalization, serious oxygen deprivation (such as following heart attack, carbon monoxide poisoning, near drowning or near suffocation), encephalitis, meningitis, or other major neurological disorder.
* History of chronic fatigue syndrome, Long-COVID.
* Other medical or psychiatric conditions that are sufficient to likely compromise current attentional function and assessment in the opinion of the investigator.
* Current ongoing treatment, deemed by the participant and their PCP as indicated for continued use during the study, with psychotropics suspected to alter attentional functioning such as antipsychotic medications, sedative hypnotics, mood stabilizers, benzodiazepines, atypical antidepressants, or anticonvulsants (listed in the Excluded Medications List, or in the opinion of the investigator are likely to interfere with study cognitive assessments).
* Participant is currently considered a suicide risk in the opinion of the Investigator, has previously made a suicide attempt, or has a prior history of, or is currently demonstrating active suicidal ideation or self-injurious behavior as measured by Columbia Suicide Severity Rating Scale at screening.
* Current treatment with guanfacine (due to the unacceptable risks of rapid withdrawal) and other medications for focus and attention problems such as Strattera, Modafinil, Armodafinil, and Clonidine that require long wash out periods (see Excluded ADHD Medications List).
* Participant plans to initiate during the primary study new concomitant prescription medications that are on the Excluded Medications List.
* Participant plans to initiate during the primary study behavioral therapy or training to improve cognition by means of game or app-based cognitive trainings or neurofeedback.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-11-23 (Actual); Study Completion 2024-11-23 (Actual)

PRIMARY OUTCOMES:
Conners Continuous Performance Task (CPT3) - HRT Std (Change from Baseline to Midpoint Mid-treatment, and Baseline to Endpoint Post-treatment) | Baseline (Day 0) and Midpoint (Day 25), and Baseline (Day 0) and Endpoint (Day 50)
  Conners CPT-HRT Std (Hit Reaction Time Standard Deviation) is the standard deviation of the reaction time of hits to target stimuli over the entire test. The calculation of the difference between Baseline and Midpoint (Mid-treatment) in the Conners HRT Std is HRT Std at Day 25 minus HRT Std at Day 0; and the difference between Baseline and Endpoint (Post-treatment) is HRT Std at Day 50 minus HRT Std at Day 0. Higher scores represent more variability in responding, reflecting poorer sustained attention control. A negative change in score represents improvement in sustained attention control.

SECONDARY OUTCOMES:
Nelson Denny Reading Comprehension Test (NDRT) - Reading Comprehension Scaled Score (Change from Baseline to Midpoint Mid-treatment, and Baseline to Endpoint Post-treatment) | Baseline (Day 0) and Midpoint (Day 25), and Baseline (Day 0) and Endpoint (Day 50)
  NDRT - Reading Comprehension Scaled Score (Reading Comp) is the total comprehension score for the full 20-minute, 36-item reading test based on the number of correct answers. The calculation of the difference between Baseline and Midpoint (Mid-treatment) in the NDRT Reading Comp is Reading Comp at Day 25 minus Reading Comp at Day 0; and the difference between Baseline and Endpoint (Post-treatment) is Reading Comp at Day 50 minus Reading Comp at Day 0. Higher scores represent more correct answer reflecting better comprehension. A positive change in score represents improvement in reading comprehension.
Barkley Adult ADHD Rating Scale (BAARS-IV) - Inattentive Subscale (Inatt). (Change from Baseline to Midpoint Mid-treatment, and Baseline to Endpoint Post-treatment) | Baseline (Day 0) and Midpoint (Day 25), and Baseline (Day 0) and Endpoint (Day 50)
  The BAARS-IV is an 18-item, self-report questionnaire for which the participant respondent rates the frequency of occurrence of ADHD symptoms and behaviors as defined by criteria outlined for ADHD in the DSM-5. Each item is scored on a 4-point scale ranging from 1 (never or rarely) to 4 (very often).
  The 18 items are grouped into 2 subscales. Each subscale produces a sub-scale score ranging from 0-36. A lower subscale score indicates less severe ADHD symptoms and behaviors.
  The calculation of the difference between Baseline and Midpoint (Mid-treatment) in the BAARS-IV Inatt score is Inatt at Day 25 minus Inatt at Day 0; and the difference between Baseline and Endpoint (Post-treatment) is Inatt at Day 50 minus Inatt at Day 0 A negative change indicates improvement on the subscale from Day 0 to Day 25 and Day 0 to Day 50.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bilder, Ph.D, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - University of California Berkeley, Berkeley, California
  - UCLA Semel Institute, Los Angeles, California